CLINICAL TRIAL: NCT06278337
Title: Etude Multicentrique Internationale rétrospective Des Patients Atteints de déficit Immunitaire associé à la moésine lié au Chromosome X (X Maid Pour X-linked Moesin Associated Immunodeficiency)
Brief Title: X-linked Moesin Associated Immunodeficiency
Acronym: X-MAIDReg
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C19-35
Record Dates: First submitted 2024-01-09; First posted 2024-02-26 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Immune Deficiency; Autoimmune Diseases; Infections; Diagnosis
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Autoimmune Diseases; Infections; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — This is an observational study involving retrospective collection of medical and biological data from X-MAID patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: genetic restrospective study — it is not an interventional study but observational

SUMMARY:
Moesin deficiency was initially described in 7 male participants aged 4 to 69 years and is characterized by lymphopenia of the 3 lineages and moderate neutropenia. Genetically, 6 out of 7 participants had the same missense mutation in the moesin gene located on the X chromosome. The 7th patient has a mutation leading to the premature introduction of a STOP codon into the protein.Clinically the 7 participants with X-linked moesin-associated immunodeficiency all presented with recurrent bacterial infections of the respiratory, gastrointestinal or urinary tracts, and some had severe varicella.Therapeutically, in the absence of a molecular diagnosis and due to his SCID-like phenotype, one patient was treated with geno-identical hematopoietic stem cell transplantation . The remaining are untreated or treated with immunoglobulin substitution and/or prophylactic antibiotics.

Since this study, the moesin gene has been integrated into DNA chips used for the molecular diagnosis of immune deficiencies in several countries. Physicians in Canada, the United States, Japan, South Africa and Europe have contacted us with a total of 16 known participants to date. Because of their very low severe, uncontrolled CMV infection and the absence of treatment recommendations, two 2 American participants were treated with allogeneic transplantation with severe post-transplant complications (1), and one of the participants died as a result of the transplant. Management of XMAID participants therefore varies widely from country to country, depending on age at diagnosis and clinical picture. It ranges from no treatment treatment (associated with recurrent infections and skin manifestations), IgIv substitution and/or antibiotic prophylaxis antibiotic prophylaxis, with low toxicity and apparent efficacy, and allogeneic transplantation, with all the risks risks involved (graft-related toxicity, graft versus host, disease, rejection, risk of infection). The Investigators therefore feel it is important to review the diagnosis, clinical presentation and management of X-MAID participants. The study the investigator propose will enable to understand the presentation of X-MAID participants, establish guidelines and provide the best treatment for each patient according to his or her clinical picture

DETAILED DESCRIPTION:
Since this study, the moesin gene has been integrated into DNA chips used for the molecular diagnosis of immune deficiencies in several countries. Physicians in Canada, the United States, Japan, South Africa and Europe have contacted us with a total of 16 known participants to date. Because of their very low severe, uncontrolled CMV infection and the absence of treatment recommendations, two 2 American participants were treated with allogeneic transplantation with severe post-transplant complications (1), and one of the participants died as a result of the transplant. Management of XMAID participants therefore varies widely from country to country, depending on age at diagnosis and clinical picture. It ranges from no treatment treatment (associated with recurrent infections and skin manifestations), IgIv substitution and/or antibiotic prophylaxis antibiotic prophylaxis, with low toxicity and apparent efficacy, and allogeneic transplantation, with all the risks risks involved (graft-related toxicity, graft versus host, disease, rejection, risk of infection). The investigators therefore feel it is important to review the diagnosis, clinical presentation and management of X-MAID participants. The study the investigators propose will enable to understand the presentation of X-MAID participants, establish guidelines and provide the best treatment for each participant according to his or her clinical picture

ELIGIBILITY:
Inclusion Criteria:

* Male patient with a mutation in the MOESIN gene (MSN)
* No objection to the collection of personal health data

Exclusion Criteria:

-

Ages: 4 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The participants are male patients (children or adults) with a mutation in the MOESIN gene (MSN) associated with an immune deficiency, regularly monitored in hospital centers because only male patients are affected by this disease, which is linked to a mutation of a gene on the X chromosome. This will enable us to determine whether symptoms and responses to treatment differ according to mutation.
  The disease can be diagnosed in the first year of life. Patients are therefore either children or adults.
Study Population: Given the small number of participants and the purpose of the study, the group may include deceased patients (at least 1 of the 16 participants). The sample size is 16 patients already identified, and possibly other patients who may be identified once the existence of the the existence of the international registry. Final enrolment will correspond to all X-MAID patients diagnosed worldwide who agree to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2026-08-12 (Estimated); Study Completion 2027-01-12 (Estimated)

PRIMARY OUTCOMES:
The main objective | through study completion, and average 3 years
  The main objective is to study the clinical results of the different therapeutic options applied to X-MAID patients, and to investigate whether there is a correlation between treatment responses and mutation position

SECONDARY OUTCOMES:
Secondary objectives1 | through study completion, and average 3 years
  Circumstances of genetic diagnosis: at what age are these patients diagnosed, and by what means? (role of prenatal screening).

OTHER OUTCOMES:
secondary objectives 2 | through study completion, and average 3 years
  What is the state of their immune system and, depending on this state, the CID or SCID classification of the disease.
secondary objective 3 | All the patients are male. As a result of their immune deficiency, patients suffer from recurrent bacterial infections of the respiratory, digestive and urinary tracts, as well as, in some cases, skin manifestations such as eczema, alopecia and molluscum
  What are the clinical manifestations of the disease (cutaneous, infectious, autoimmune)?
secondary objectives 4 | Among patients diagnosed in the first years of life, none showed developmental defects.
  What impact does the disease have on their development?
secondary objective 5 | Treatments range from no prophylaxis at all to antibiotic prophylaxis, with or without immunoglobulin therapy, granulocyte-colony-stimulating factor therapy or hematopoietic stem cell allograft.
  What are the treatments and their consequences?

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle ANDRE, doctor, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (10):
- United States (3):
  - National Institutes of Health, Bethesda, Maryland
  - Perelman School of medecine, Philadelphia, Pennsylvania
  - Brown University, Providence, Rhode Island
- Genomic Research Centre, School of Biomedical Sciences Institute of Health and Biomedical Innovation, Brisbane, Australia
- Hôpital Universitaire de la Reine Fabiola, Brussels, Belgium
- France (3):
  - Hôpital Necker, Paris, PARIS
  - CHU Rennes, CNRS UMR 629, Rennes
  - CHU St Etienne Hôpital Nord, Saint-Etienne
- Tokyo Medical and Dental University (TMDU), Bunkyō City, Japan
- Departments of Internal Medicine and Immunology, Rotterdam, Netherlands